CLINICAL TRIAL: NCT00576719
Title: Intensive Treatment of Adolescent Panic and Agoraphobia
Brief Title: Effectiveness of Intensive Cognitive Behavioral Therapy in Treating Adolescent Panic Disorder and Agoraphobia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH068277 (NIH); R01MH068277 (NIH); DSIR 84-CTS
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Panic Disorder; Agoraphobia
MeSH Terms: conditions — Panic Disorder; Agoraphobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive intensive cognitive behavioral therapy treatment without parent involvement
  Interventions: Behavioral: Intensive panic control treatment without parent involvement
- 2 (Experimental): Participants will receive intensive cognitive behavioral therapy treatment with parent involvement
  Interventions: Behavioral: Intensive panic control treatment with parent involvement
- 3 (Placebo Comparator): Waitlist control group
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: Intensive panic control treatment without parent involvement — Intensive panic control treatment without parent involvement is an 8-day, intensive form of cognitive behavioral therapy (CBT) with exposure, including 15-20 hours of direct therapist contact. The basic treatment components are psychoeducation about anxiety, restructuring anxiety-provoking thoughts, exposure to bodily sensations that trigger panic, and in vivo exposures.
  Arms: 1
Behavioral: Intensive panic control treatment with parent involvement — Intensive panic control treatment with parent involvement involves the same form of intensive CBT, but with direct parent involvement. Parents will attend the last 30 minutes of didactic sessions, complete homework assignments, learn ways to coach their children, and participate in selected exposures.
  Arms: 2
Other: Waitlist control — Waitlist control participants will receive active treatment (treatment with or without family involvement) after 6 weeks of waitlist.
  Arms: 3

SUMMARY:
This study will evaluate the effectiveness of intensive cognitive behavioral therapy in treating adolescents with panic disorder with agoraphobia.

DETAILED DESCRIPTION:
Panic disorder (PD) in adolescents is a prevalent and chronic anxiety disorder. People with PD experience unexpected attacks of fear, along with elevated heart rate, dizziness, faintness, weakness, and increased sweating. During these panic attacks, people may feel numbness in their hands, flushed or chilled, nauseous, or pain in the chest, and they may lose touch with reality. PD can lead to substantial social impairment for adolescents, including avoidance of school, independent activities, and peer involvement. When PD progresses so far that a person avoids public places where a panic attack might occur, the person is said to have a condition known as agoraphobia. Weekly sessions of cognitive behavioral therapy (CBT) appear to be effective in treating panic disorder with agoraphobia (PDA). However, many adolescents with PDA and their families report the need for a more immediate relief from the disorder. This study will evaluate the effectiveness of intensive CBT in treating adolescents with PDA.

Participants in this single blind study will be randomly assigned to one of three conditions: intensive CBT treatment including family members, intensive CBT treatment without family members, or a waitlist control group. All participants in the intensive CBT treatment groups will undergo 8 days of intensive CBT, for a total of 6 sessions. On Days 1 through 3 of treatment, participants will attend daily, 2-hour CBT sessions. The CBT sessions will include psychoeducation about anxiety, tactics to restructure anxiety-provoking thoughts, and exposure to bodily sensations that trigger panic. On Days 4 and 5, participants will meet with a therapist to learn ways to approach previously feared situations. On Days 6 and 7, participants will continue working independently or with family members to solidify skills. On Day 8, participants will attend a final 2-hour session to consolidate skills, review the independent weekend activities, and discuss ways to apply skills to the home environment. Parents of participants in the parental involvement group will attend the last 30 minutes of sessions, complete homework assignments, learn ways to coach their children through episodes, and participate in selected exposures. After 6 weeks of waitlist, participants in the waitlist control group will receive active treatment following the same procedures as the initial active treatment. All participants will be assessed at Months 3, 6, and 12 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for principal diagnosis of PD or PDA prior to treatment
* Adolescent must be accompanied by at least one parent or caregiver
* If on medication, there must be a 1-month stabilization period for benzodiazepines or 3-month stabilization period for SSRIs or tricyclics prior to study entry

Exclusion Criteria:

* Positive diagnosis of schizophrenia, pervasive developmental disorder, organic brain syndrome, mental retardation, or current suicidal ideation
* Unavailability of at least one parent or caregiver
* Refusal of parent to accept random assignment to treatment condition
* Refusal of parent or adolescent to accept stabilization of medication
* Adolescent with parent who has any condition that would limit ability to understand treatment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2005-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule-Child and Parent Versions: Clinical Severity Rating, Agoraphobia Ratings, Panic Attack Frequency Scores, and Internal Sensation Anxiety Ratings | Measured at Months 3, 6, and 12 post-treatment
Panic Disorder Severity Scale-Child Version | Measured at Months 3, 6, and 12 post-treatment

SECONDARY OUTCOMES:
Multidimensional Anxiety Scale for Children | Measured at Months 3, 6, and 12 post-treatment
Childhood Anxiety Sensitivity Index | Measured at Months 3, 6, and 12 post-treatment
Fear and Avoidance Hierarchy | Measured at Months 3, 6, and 12 post-treatment
Children's Depression Inventory | Measured at Months 3, 6, and 12 post-treatment
The Panic Attack Record | Measured at Months 3, 6, and 12 post-treatment
Subjective Symptoms Scale | Measured at Months 3, 6, and 12 post-treatment
Panic and Phobia Questionnaire | Measured at Months 3, 6, and 12 post-treatment
Participant Global Impression of Improvement (PGI) | Measured at Months 3, 6, and 12 post-treatment
Perceptions of Treatment Questionnaire: Adolescent and Parent Versions | Measured at Months 3, 6, and 12 post-treatment
Children's Perception Scale (Locus of Control Scale) | Measured at Months 3, 6, and 12 post-treatment
Child Behavior Checklist (CBCL) | Measured at Months 3, 6, and 12 post-treatment
Stress Index for Parents of Adolescents | Measured at Months 3, 6, and 12 post-treatment
Parenting Locus of Control Scale | Measured at Months 3, 6, and 12 post-treatment
Therapy Attitude Inventory | Measured at Months 3, 6, and 12 post-treatment
Family Assessment Measure (FAM) | Measured at Months 3, 6, and 12 post-treatment
Depression Anxiety and Stress Scale (DASS) | Measured at Months 3, 6, and 12 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Donna Pincus, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States